CLINICAL TRIAL: NCT04579575
Title: Added Value of Ovarian-Adnexal Reporting and Data System in Evaluation of Ovarian Lesions
Brief Title: Added Value of O-RADS in Evaluation of Ovarian Lesions
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdel Maged Mohamed, Principal investigator, Assiut University
Other Study IDs: O-RADS value in ovarian lesion
Record Dates: First submitted 2020-09-23; First posted 2020-10-08 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Ovarian Diseases
MeSH Terms: conditions — Ovarian Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Trans-abdominal Ultrasound — All patients will undergo trans- abdominal and trans-vaginal examination (The trans-abdominal US was performed for virgin patients or patients with large tumors that cannot be completely seen by the TV route) performed on the devices available in South Egypt Cancer Institute in supine position.
  The most important b-mode parameters (such as gain, frequency, number of foci and their depth, etc.) of the US machines were manually adjusted to obtain similar image impressions.
  * The morphological features of each AM, and independently categorized the US images of each AM according to the O-RADS published by ACR and GI-RADS simple rules . The results of consensus reviewing were used to calculate the validity of each US classification system.
  * The definite diagnoses of AM were preferentially established based on
  Histo-pathological findings and other modalities.
  Other Names: Trans-vaginal Ultrasound

SUMMARY:
To detect added value of O-RADS in evaluation of ovarian lesions and compare O-RADS with GI-RADS regarding malignancy rate, the validity and reliability through pathological results and other modalities

DETAILED DESCRIPTION:
Ultrasound (US) continues to be the initial imaging modality of choice for the identification and characterization of adnexal masses (AM) . Structured reporting of AM findings was identified by a Society of Radiologists in Ultrasound consensus working group as a target for the investigation to improve the management of women with AM .

Many established guidelines and structured reporting have been developed using sonography to characterize AM, including subjective assessment, simple scoring systems, and statistically derived scoring systems .

In 2008, the International Ovarian Tumor Analysis (IOTA) group proposed the use of US simple rules for the diagnosis of ovarian malignancy. These are based on a set of five US features indicative for a benign tumor (B features), and five US features indicative for a malignant tumor (M features)

. In 2009, the Gynecology Imaging Reporting and Data System (GI-RADS) was designed as an attempt allowing standardized reporting of AM. This system is based on recognition patterns and criteria provided by the IOTA.

The American College of Radiology (ACR) published the Ovarian-Adnexal Reporting and Data System (O-RADS), which provides an up-to-date suggestion to stratify the AM according to sonographic features. The O-RADS offers a comprehensive algorithm that categorizes AM by their possibility of being normal (O-RADS 1), to high risk of malignancy (O-RADS 5) .

For the application of the US classification system of AM in clinical settings, it is essential to evaluate their validity and reproducibility. Several studies have investigated the validity of these risk stratification systems in the assessment of AM. However, data on the comparability and reproducibility of the systems are limited.

The purpose of this study is To detect added value of O-RADS in evaluation of ovarian lesions and compare O-RADS with GI-RADS regarding malignancy rate , the validity and reliability through pathological results.

ELIGIBILITY:
Inclusion Criteria:

* All newly diagnosed patients with ovarian lesions referred to the radiology department.
* Must be able to be examined.

Exclusion Criteria:

* Patients younger than 17 years old
* Patient who refused to be a part of the study and undergo examination.

Ages: 17 Years to 75 Years | Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ovarian lesions expected to visit Radiology Department at South Egypt Cancer Institute or Assiut University Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-12-20 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Added value of Ovarian-Adnexal Reporting and Data System in evaluation of 30 participants with ovarian lesions regarding malignancy rate ,the validity and reliability after comparison with pathology specimens results . | Baseline
  Evaluation of the ovarian lesions by Trans-abdominal and Trans-vaginal Ultrasound for diagnosis of ovarian malignancy as early as possible for further management

CONTACTS AND LOCATIONS:
Overall Officials: Hisham Moustafa Kamel, Study Director — Assiut University; Haisam Ahmed Samy Aly Atta, Study Director — South Egypt Cancer Institute ,Assiut University; Doaa Mohamed Fouad, Study Director — South Egypt Cancer Institute ,Assiut University

REFERENCES:
- [Background] Liu J, Xu Y, Wang J. Ultrasonography, computed tomography and magnetic resonance imaging for diagnosis of ovarian carcinoma. Eur J Radiol. 2007 Jun;62(3):328-34. doi: 10.1016/j.ejrad.2007.02.040. Epub 2007 Apr 11. PMID 17433597
- [Background] Levine D, Brown DL, Andreotti RF, Benacerraf B, Benson CB, Brewster WR, Coleman B, DePriest P, Doubilet PM, Goldstein SR, Hamper UM, Hecht JL, Horrow M, Hur HC, Marnach M, Patel MD, Platt LD, Puscheck E, Smith-Bindman R; Society of Radiologists in Ultrasound. Management of asymptomatic ovarian and other adnexal cysts imaged at US Society of Radiologists in Ultrasound consensus conference statement. Ultrasound Q. 2010 Sep;26(3):121-31. doi: 10.1097/RUQ.0b013e3181f09099. PMID 20823748
- [Background] Timmerman D, Valentin L, Bourne TH, Collins WP, Verrelst H, Vergote I; International Ovarian Tumor Analysis (IOTA) Group. Terms, definitions and measurements to describe the sonographic features of adnexal tumors: a consensus opinion from the International Ovarian Tumor Analysis (IOTA) Group. Ultrasound Obstet Gynecol. 2000 Oct;16(5):500-5. doi: 10.1046/j.1469-0705.2000.00287.x. No abstract available. PMID 11169340
- [Background] Timmerman D, Van Calster B, Testa A, Savelli L, Fischerova D, Froyman W, Wynants L, Van Holsbeke C, Epstein E, Franchi D, Kaijser J, Czekierdowski A, Guerriero S, Fruscio R, Leone FPG, Rossi A, Landolfo C, Vergote I, Bourne T, Valentin L. Predicting the risk of malignancy in adnexal masses based on the Simple Rules from the International Ovarian Tumor Analysis group. Am J Obstet Gynecol. 2016 Apr;214(4):424-437. doi: 10.1016/j.ajog.2016.01.007. Epub 2016 Jan 19. PMID 26800772
- [Background] Van Calster B, Van Hoorde K, Valentin L, Testa AC, Fischerova D, Van Holsbeke C, Savelli L, Franchi D, Epstein E, Kaijser J, Van Belle V, Czekierdowski A, Guerriero S, Fruscio R, Lanzani C, Scala F, Bourne T, Timmerman D; International Ovarian Tumour Analysis Group. Evaluating the risk of ovarian cancer before surgery using the ADNEX model to differentiate between benign, borderline, early and advanced stage invasive, and secondary metastatic tumours: prospective multicentre diagnostic study. BMJ. 2014 Oct 15;349:g5920. doi: 10.1136/bmj.g5920. PMID 25320247
- [Background] Van Calster B, Timmerman D, Valentin L, McIndoe A, Ghaem-Maghami S, Testa AC, Vergote I, Bourne T. Triaging women with ovarian masses for surgery: observational diagnostic study to compare RCOG guidelines with an International Ovarian Tumour Analysis (IOTA) group protocol. BJOG. 2012 May;119(6):662-71. doi: 10.1111/j.1471-0528.2012.03297.x. Epub 2012 Mar 6. PMID 22390753
- [Background] Amor F, Vaccaro H, Alcazar JL, Leon M, Craig JM, Martinez J. Gynecologic imaging reporting and data system: a new proposal for classifying adnexal masses on the basis of sonographic findings. J Ultrasound Med. 2009 Mar;28(3):285-91. doi: 10.7863/jum.2009.28.3.285. PMID 19244063
- [Background] Amor F, Alcazar JL, Vaccaro H, Leon M, Iturra A. GI-RADS reporting system for ultrasound evaluation of adnexal masses in clinical practice: a prospective multicenter study. Ultrasound Obstet Gynecol. 2011 Oct;38(4):450-5. doi: 10.1002/uog.9012. PMID 21465605
- [Background] Kaijser J, Sayasneh A, Van Hoorde K, Ghaem-Maghami S, Bourne T, Timmerman D, Van Calster B. Presurgical diagnosis of adnexal tumours using mathematical models and scoring systems: a systematic review and meta-analysis. Hum Reprod Update. 2014 May-Jun;20(3):449-62. doi: 10.1093/humupd/dmt059. Epub 2013 Dec 9. PMID 24327552
- [Background] Andreotti RF, Timmerman D, Benacerraf BR, Bennett GL, Bourne T, Brown DL, Coleman BG, Frates MC, Froyman W, Goldstein SR, Hamper UM, Horrow MM, Hernanz-Schulman M, Reinhold C, Strachowski LM, Glanc P. Ovarian-Adnexal Reporting Lexicon for Ultrasound: A White Paper of the ACR Ovarian-Adnexal Reporting and Data System Committee. J Am Coll Radiol. 2018 Oct;15(10):1415-1429. doi: 10.1016/j.jacr.2018.07.004. Epub 2018 Aug 24. PMID 30149950
- [Background] Andreotti RF, Timmerman D, Strachowski LM, Froyman W, Benacerraf BR, Bennett GL, Bourne T, Brown DL, Coleman BG, Frates MC, Goldstein SR, Hamper UM, Horrow MM, Hernanz-Schulman M, Reinhold C, Rose SL, Whitcomb BP, Wolfman WL, Glanc P. O-RADS US Risk Stratification and Management System: A Consensus Guideline from the ACR Ovarian-Adnexal Reporting and Data System Committee. Radiology. 2020 Jan;294(1):168-185. doi: 10.1148/radiol.2019191150. Epub 2019 Nov 5. PMID 31687921